CLINICAL TRIAL: NCT06040736
Title: Point-of-care Ultrasound to Assess Hydronephrosis in Patients Presenting With Acute Kidney Injury in the Emergency Department: a Prospective Comparative Pragmatic Study
Brief Title: Point-of-care Ultrasound to Assess Hydronephrosis in Patients With Acute Kidney Injury in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0158
Record Dates: First submitted 2023-09-04; First posted 2023-09-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury; Urinary Tract Obstruction
Keywords: Point-of-care ultrasound; Acute kidney injury; Hydronephrosis; urinary tract obstruction; Emergency Medicine
MeSH Terms: conditions — Acute Kidney Injury; Hydronephrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with acute kidney injury: Emergency department patients presenting with acute kidney injury, regardless of their complaint for ED admission. AKI is defined based on increase in serum creatinine (SCr) levels according to Kdigo criteria Patients will undergo both a bedside point of care ultrasonography and a central radiology imaging evaluation of hydronephrosis as part of routine care

SUMMARY:
Acute kidney injury (AKI) is a common diagnosis in the emergency department (ED), and urinary tract obstruction is a contributing cause that requires rapid diagnosis and therapeutic management. This observational study aims at assessing the accuracy of point-of-care ultrasound (POCUS), performed by the emergency physician (EP) for the detection of dilatation or distension of the kidney secondary to urinary tract obstruction, in emergency department patients presenting with acute kidney injury (AKI). Participants will undergo a bedside POCUS of the urinary tract by the EP followed by central imaging evaluation by a radiologist (either ultrasound or renal computed tomography (CT) or both). Researchers will compare both diagnosis. Study hypothesis is that trained emergency physicians can rapidly and reliably diagnose renal tract obstruction at POCUS in the context of AKI.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common diagnosis in the emergency department (ED), and urinary tract obstruction is a contributing cause that requires rapid diagnosis and therapeutic management. Hydronephrosis is a dilatation or distension of the kidney secondary to urinary tract obstruction. It can be diagnosed at ultrasonography or computed tomography. Assessment of the renal tract and detection of hydronephrosis is a core component of the emergency medicine Point-of-Care Ultrasound (Pocus) curriculum. The primary objective of this study is to compare the performance of point-of-care ultrasound performed by the emergency physician to that of central radiology imaging (US or CT) by a radiologist, to diagnose hydronephrosis in patients presenting with AKI in the ED. All imaging exams will be performed as part of routine evaluation, Pocus will be carried out by a trained EP blinded from radiology imaging results.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute kidney injury defined by changes in serum creatinine (sCr) level between the index sCr at ED admission and pre and/or post sCr controls (Kidney Disease Improving Global Outcome criteria)
* Patient who does not oppose to the use of their data

Exclusion Criteria:

* Vesical globe
* Polycystic kidney disease
* Known renal tumor
* Horseshoe kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the emergency department of Montpellier university hospital
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Performance of pont of care ultrasound (POCUS) for the diagnosis of hydronephrosis | 1 day (Emergency department (ED) length of stay)
  Performance of POCUS for the detection of hydronephrosis compared to radiology imaging as the gold standard (Sensitivity, Specificity, Negative Predictive Value, Positive Predicted Value)

SECONDARY OUTCOMES:
Level of agreement between ED Pocus and central radiology imaging for the diagnosis of hydronephrosis | 1 day (ED length of stay)
  Agreement between Pocus and radiology examination (radiology ultrasound (US) or Computed Tomography (CT) for the diagnosis of hydronephrosis
Risk Factors for POCUS misdiagnosis | 1 day (ED length of stay)
  Factors associated with misdiagnosis of hydronephrosis at POCUS

CONTACTS AND LOCATIONS:
Overall Officials: Mustapha SEBBANE, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- university hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No